CLINICAL TRIAL: NCT01717950
Title: Phase 1 Study of the Safety and Immunogenicity of Na-APR-1 (M74)/Alhydrogel® in Healthy Adults
Brief Title: Safety and Immunogenicity of the Na-APR-1 Hookworm Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: George Washington University (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Sponsor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SVI-12-01
Record Dates: First submitted 2012-10-25; First posted 2012-10-31 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Hookworm Infection; Hookworm Disease
Keywords: Human Hookworm; Necator americanus; Hookworm; Hookworm Disease; Iron-deficiency anemia; Soil-transmitted helminth infection; Neglected Tropical Disease; Na-APR-1
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis; Anemia, Iron-Deficiency; Neglected Diseases | interventions — GLA-AF adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 30 µg Na-APR-1 (M74)/Alhydrogel® (Experimental)
  Interventions: Biological: Na-APR-1 (M74)/Alhydrogel®
- 30 µg Na-APR-1 (M74)/Alhydrogel® plus 2.5 µg GLA-AF (Experimental)
  Interventions: Biological: Na-APR-1 (M74)/Alhydrogel®; Biological: Gluco-Pyranosylphospho-Lipid A Aqueous Formulation
- 30 µg Na-APR-1 (M74)/Alhydrogel® plus 5.0 µg GLA-AF (Experimental)
  Interventions: Biological: Na-APR-1 (M74)/Alhydrogel®; Biological: Gluco-Pyranosylphospho-Lipid A Aqueous Formulation
- 100 µg Na-APR-1 (M74)/Alhydrogel® (Experimental)
  Interventions: Biological: Na-APR-1 (M74)/Alhydrogel®
- 100 µg Na-APR-1 (M74)/Alhydrogel® plus 2.5 µg GLA-AF (Experimental)
  Interventions: Biological: Na-APR-1 (M74)/Alhydrogel®; Biological: Gluco-Pyranosylphospho-Lipid A Aqueous Formulation
- 100 µg Na-APR-1 (M74)/Alhydrogel® plus 5.0 µg GLA-AF (Experimental)
  Interventions: Biological: Na-APR-1 (M74)/Alhydrogel®; Biological: Gluco-Pyranosylphospho-Lipid A Aqueous Formulation

INTERVENTIONS:
Biological: Na-APR-1 (M74)/Alhydrogel® — The Na-APR-1 (M74) candidate vaccine contains the recombinant Na-APR-1 (M74) protein expressed by Nicotiana plants. Purified Na-APR-1 (M74) was subsequently adsorbed onto aluminum hydroxide gel (Alhydrogel®) and suspended in a solution containing 10 mM imidazole, 150 mM sodium chloride and 0.3% Empigen BB, with pH 7.4 ± 0.1. The final concentration of Na-APR-1 (M74) in the drug product is 0.1 mg/ml, whereas that of Alhydrogel® is 0.8 mg/ml. Different doses of Na-APR-1 (M74) will be delivered by injecting different volumes of the 0.1 mg/ml Na-APR-1 (M74) preparation.
  Other Names: Na-APR-1; Necator americanus Aspartic Protease-1
Biological: Gluco-Pyranosylphospho-Lipid A Aqueous Formulation — GLA-AF contains a synthetic monophosphoryl lipid A (MPL) molecule that has Toll-Like Receptor-4 agonist activity. MPL is itself derived from the lipopolysaccharide (LPS) of Salmonella minnesota, a natural TLR4 agonist that is pyrogenic and can induce toxic shock. LPS, and more specifically, its lipid A component, has long been known for its strong adjuvant effects; however, its high toxicity has precluded its use in a vaccine formulation.
  Other Names: GLA-AF
  Arms: 100 µg Na-APR-1 (M74)/Alhydrogel® plus 2.5 µg GLA-AF; 100 µg Na-APR-1 (M74)/Alhydrogel® plus 5.0 µg GLA-AF; 30 µg Na-APR-1 (M74)/Alhydrogel® plus 2.5 µg GLA-AF; 30 µg Na-APR-1 (M74)/Alhydrogel® plus 5.0 µg GLA-AF

SUMMARY:
Hookworms digest hemoglobin from erythrocytes for use as an energy source via a proteolytic cascade that begins with the aspartic protease, APR-1. Vaccination with recombinant APR-1 has protected animals from infection in challenge studies. This study will evaluate the safety and immunogenicity of two formulations of Na-APR-1 (M74) in healthy adult volunteers when co-administered with different concentrations of the immunostimulant GLA-AF.

DETAILED DESCRIPTION:
Open-label, dose-escalation phase 1 clinical trial in healthy, hookworm-naïve adults:

* Study site: George Washington Medical Faculty Associates, Washington, DC
* Number of participants: 40 in 2 cohorts of 20.

In Cohort 1 five (5) volunteers will receive 30 µg Na-APR-1 (M74) /Alhydrogel®, five (5) will receive 30 µg Na-APR-1 (M74)/Alhydrogel® plus 2.5 µg GLA-AF, and ten (10) will receive 30 µg Na-APR-1 (M74) /Alhydrogel® plus 5 µg GLA-AF. In Cohort 2 five (5) volunteers will receive 100 µg Na-APR-1 (M74)/Alhydrogel®, five (5) will receive 100 µg Na-APR-1 (M74) /Alhydrogel® plus 2.5 µg GLA-AF, and ten (10) will receive 100 µg Na-APR-1 (M74)/Alhydrogel® plus 5 µg GLA-AF.

The cohorts will be enrolled in a staggered fashion with safety data assessed prior to the Na-APR-1 dose escalation from 30 to 100 µg. In addition, within each cohort, vaccinations will be staggered such that formulations containing 0, 2.5, and 5 µg GLA-AF will be tested sequentially: for example, those receiving Na-APR-1 (M74)/Alhydrogel® in combination with 2.5 µg GLA-AF will be vaccinated no sooner than 3 days after the last volunteer is vaccinated with the formulation containing no GLA-AF, whereas those vaccinated with Na-APR-1 (M74)/Alhydrogel® plus 5 µg GLA-AF will be vaccinated no sooner than 7 days after the last one receives the 2.5 µg GLA-AF formulation.

* Immunization schedule: Study days 0, 56 and 112.
* Route: IM in the deltoid muscle.
* Doses of Na-APR-1 (M74) to be tested: 30 and 100 µg.
* Doses of Alhydrogel®: 240 and 800 µg for the 30 and 100 µg doses of Na-APR-1 (M74), respectively.
* Doses of GLA-AF to be tested: 2.5 µg and 5 µg.
* Study duration: 44 weeks (10 months) per study participant; total duration of the study estimated at approximately 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 50 years, inclusive.
* Good general health as determined by means of the screening procedure.
* Available for the duration of the trial (44 weeks).
* Willingness to participate in the study as evidenced by signing the informed consent document.

Exclusion Criteria:

* Pregnancy as determined by a positive urine human choriogonadotropin (hCG) (if female).
* Participant unwilling to use reliable contraception methods up until one month following the third immunization (if female and not surgically sterile, abstinent or at least 2 years post-menopausal).
* Currently lactating and breast-feeding (if female).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
* Known or suspected immunodeficiency.
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
* Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than trace protein or blood on urine dipstick testing).
* Laboratory evidence of hematologic disease (hemoglobin <11.5 g/dl [females] or <12.5 g/dl [males]; absolute leukocyte count <3600/mm3 or >10.7 x 103/mm3; absolute neutrophil count [ANC] <1700/ mm3; absolute lymphocyte count <700/mm3; or platelet count <140,000/mm3).
* Laboratory evidence of a coagulopathy (PTT or PT INR greater than 1.1-times the upper reference limit).
* Serum glucose (random) greater than 1.2-times the upper reference limit.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Participation in another investigational vaccine or drug trial within 30 days of starting this study.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma as defined by the need for daily use of inhalers or emergency clinic visit or hospitalization within 6 months of the volunteer's expected first vaccination in the study.
* Positive ELISA for hepatitis B surface antigen (HBsAg).
* Positive confirmatory test for HIV infection.
* Positive confirmatory test for hepatitis C virus (HCV) infection.
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of the volunteer's expected first vaccination in this study.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to the volunteer's expected first vaccination in the study.
* History of a surgical splenectomy.
* Receipt of blood products within the past 6 months.
* History of previous infection with hookworm or residence for more than 6 months in a hookworm-endemic area.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Vaccine-related Adverse Events | Day 290
  The frequency of immediate, systemic, and local injection site adverse events will be summarized. Adverse events will be assessed by study team members at 1 hour post-vaccination as well as 3, 7, 14, and 28 days following each vaccination. In addition, study participants will be asked to complete symptom diaries for the 7 days after each vaccination.

SECONDARY OUTCOMES:
IgG antibody response to Na-APR-1 | 14 days after final vaccination
  Dose and formulation of Na-APR-1 that generates the highest IgG antibody response at Day 126 (14 days after final vaccination), as determined by an indirect enzyme-linked immunosorbent assay (ELISA).
B cell response to Na-APR-1 | Study Days 14, 70, 126, 140 and 290
  Dose and formulation of the Na-APR-1 (M74) vaccine that results in the highest production of Na-APR-1 (M74) specific B cells and subtypes (memory or plasma).
Exploratory cellular immune response to Na-APR-1 | Study Days 14, 70, 126, 140 and 290
  Exploratory studies of the cellular immune responses to the Na APR-1 (M74) antigen both before and after immunization.

CONTACTS AND LOCATIONS:
Overall Officials: David J Diemert, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

REFERENCES:
- Available data/document: Clinical Study Report — https://smhs.gwu.edu/mitm-crg/